CLINICAL TRIAL: NCT05005858
Title: Modified Ridge Splitting Technique Using Autogenous Bone Blocks (MRS)
Acronym: MRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Collaborators: NSK Europe GmbH (Industry); Hungarian Dental Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52158-2/2015/EKU
Record Dates: First submitted 2021-06-04; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-06

CONDITIONS: Alveolar Bone Resorption; Alveolar Ridge Enlargement

STUDY DESIGN:
Intervention Model Description: * Procedure: alveolar ridge splitting
  * Procedure: bone core biopsy After 3 month healing time reentry took place and bone core biopsy samples were collected from the augmented bone of the maxillary sinuses with a trephine drill. Biopsy samples were collected from the sites where the dental implants were to be placed.
  * Device: dental implant placement During reentry after bone biopsy dental implants were placed.
  * Clinical measurements:
  Measurements were carried out using Williams probe
  * Histomorphometric measurements
  * Micro-CT analysis
Masking Description: The specialis tasked with histomorphometric, micro-CT analysis has no knowledge on the intervention method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autograft (Experimental): The filler used in ridge splitting is autologous bone block harvested from mandible
  * Interventions:
  * Procedure: ridge splitting
  * Procedure: bone core biopsy
  * Device: dental implant placement
  * Measurement: clinical measurement with Williams probe
  * Micro-CT analysis
  * Histomorphometric measurements
  Interventions: Procedure: Alveolar ridge splitting; Device: Creating osteotomies with piezoelectric device

INTERVENTIONS:
Procedure: Alveolar ridge splitting — Patients with Kennedy Class I. and II. mandibles with insufficient bone width were included in this study. Ridge splitting was carried out with the use of a piezoelectric surgery device by preparing osteotomies and after mobilization of the buccal cortical by placing an autologous bone block harvested from the retromolar region as a spacer between the buccal and lingual cortical plates. Block-grafts were stabilized by osteosynthesis screws. Implant placement was carried out after a 3-month healing period.
Device: Creating osteotomies with piezoelectric device — Osteotomies were carried out with piezoelectric surgery device (NSK Variosurg3 Ultrasonic Bone Surgery System, NSK Europe GmbH, Eschborn, Germany)

SUMMARY:
In this clinical study ridge splitting procedures are preformed using autogenous bone blocks. After a 3-month healing, at the time of dental implant placement bone core biopsy samples are harvested. The samples undergo micro-Ct and histomorphometric analysis.

DETAILED DESCRIPTION:
Patients were required to rinse with a 0.2% chlorhexidine solution for 1 min before surgery. Under local anesthesia, a full-thickness flap was raised from a crestal incision with a mesial releasing incision to access the alveolar ridge and the retromolar area. A midcrestal osteotomy was preformed, leaving a safety zone of at least 2 mm from the adjacent tooth. Two vertical releasing osteotomies were performed at the mesial and distal ends of the mid-crestal osteotomy. Apically, the vertical osteotomies were connected horizontally with a superficial corticotomy. Osteotomies and corticotomies were carried out using a piezoelectronic device (NSK Variosurg3 Ultrasonic Bone Surgery System, NSK Europe GmbH, Eschborn, Germany.) Chisels were inserted in the midcrestal osteotomy to create a green-stick fracture to allow extensive mobilization of the buccal cortical.

After mobilization of the buccal cortical, an autologous bone block with dimensions corresponding to that of the bone defect created in the recipient site was harvested from the retromolar area and was placed as a spacer between the buccal and lingual cortical plates. The block was stabilized using osteosynthesis screws (Meisinger Screw System, Hager and Meisinger GmbH, Neuss, Germany). Both lingual and buccal flaps were mobilized to allow tension-free primary closure. The flap was closed with horizontal mattress sutures, and then single interrupted sutures closed the edges of the flaps. Suture removal took place after 14 days. All patients received amoxicillin and clavulanate (Aktil Duo 875 mg/125 mg, Sandoz Hungária Kft., Budapest, Hungary) 1 g twice per day, starting at the day of the surgery and continuing for 7 days. In case of amoxicillin allergy, clindamycin (Dalacin 300 mg, Pfizer Inc., New York, NY, USA) was prescribed four times a day for 7 days. Furthermore, a non-steroid anti-inflammatory drug, diclofenac (Cataflam 50 mg, Novartis Hungária Kft., Budapest, Hungary), 3 times a day for 3 days, and 0.2% chlorhexidine mouth rinse (Corsodyl, GlaxoSmithKline Consumer Healthcare GmbH & Co. KG, München, Germany), twice a day for 2 weeks, were prescribed to the patients. During the healing period, patients did not wear temporary prostheses.

Surgical re-entry took place after 3 months of healing. Implant bed preparation was carried out with rotatory instruments powered by a surgical micromotor (MasterSurg Surgical Systems, KaVo Dental Systems Japan, Co., Ltd., Tokyo, Japan). A trephine drill with an external diameter of 3.0 mm and an internal diameter of 2.0 mm (330 205 486 001 020 Hager and Meisinger GmbH, Neuss, Germany) with external cooling at a drill rotation speed of 800 rpm to the depth of 8 mm was used to remove bone core biopsy samples for histologic analysis. Implant beds were finalized according to the instructions of the implant manufacturer at a rotation speed of 800 rpm. Implants (Nobel Replace Conical Connection, Nobel Biocare AG, Kloten, Switzerland) were placed submerged in the augmented bone. Implant uncovery procedure took place 3 months after implant placement.

Clinical measurements:

Measurements were carried out using Williams probe (Karl Hammacher GmbH, Solingen, Germany) prior to ridge splitting surgery after the full thickness flap elevation, to evaluate the width of the alveolar ridge (preoperative measurement) and after a 3-month healing period, before implant placement (postoperative measurement). The width of the alveolar ridges was measured at 3, 10, and 15 mm from the reference point.

Histomorphometry:

Bone core biopsy material was fixed in 10% buffered formaldehyde solution. Following decalcination and dehydration, the biopsy material was embedded in paraffin and 20 µm sections were prepared. The sections were stained with routine haematoxylin eosin stain. Sections were evaluated under a light microscope in magnification 40×-400× .

Micro-CT analysis:

The bone core biopsy samples were scanned using a microcomputed tomography (μCT) scanner (Skyscan 1172 X-ray microtomograph, Bruker µCT, Kontich, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Mandibular ridge width at least 3 mm;
* Ridge height at least 11 mm;
* Spongiosa between the two cortical plates at least 1 mm

Exclusion Criteria:

* History of uncontrolled medical disorders;
* History of systemic diseases or medication that alter bone metabolism;
* Poor oral hygiene;
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical measurements | After the 3-month healing period, at the implant placement.
  Clinical measurements were carried out using Williams probe (Karl Hammacher GmbH, Solingen, Germany) prior to ridge splitting surgery after the full thickness flap elevation, to evaluate the width of the alveolar ridge (preoperative measurement) and after a 3-month healing period, before implant placement (postoperative measurement). The width of the alveolar ridges was measured at 3, 10, and 15 mm from the reference point, which was the distal marginal bone of the last tooth of the quadrant. To ensure that preoperative and postoperative measurement sites corresponded, we placed the tip of the Williams probe on the reference point described and the markings of the probe to the highest ridge of the lingual cortical.
BV/TV bone volume fraction | After the 3-month healing period
  Bone volume compared to total volume in micro-CT reconstruction

SECONDARY OUTCOMES:
Newly formed bone percentage | After the 3-month healing period
  Newly formed bone area compared to total area in histomorphometry

CONTACTS AND LOCATIONS:
Overall Officials: Márton Kivovics, Ph.D, Study Director — Semmelweis University
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Penzes D, Simon F, Mijiritsky E, Nemeth O, Kivovics M. A Modified Ridge Splitting Technique Using Autogenous Bone Blocks-A Case Series. Materials (Basel). 2020 Sep 11;13(18):4036. doi: 10.3390/ma13184036. PMID 32932942